CLINICAL TRIAL: NCT02377986
Title: Augmenting Buried in Treasures Workshop (BIT) With In-home Decluttering Practice for Individuals With Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Carolyn I. Rodriguez, Associate Chair for Inclusion and Diversity, Department of Psychiatry, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7073
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: BIT+In-home Decluttering (Experimental): Patients who have not received the BIT workshop through our previous study (IRB 6681) will receive BIT+in-home decluttering practice.
  Interventions: Behavioral: BIT+in-home decluterring; Behavioral: In-Home Decluttering

INTERVENTIONS:
Behavioral: BIT+in-home decluterring — BIT Workshop + In-home decluttering practice
Behavioral: In-Home Decluttering — In-home decluttering practice

SUMMARY:
Patients participate in Buried in Treasures Workshop (BIT) that has been shown to improve symptoms of hoarding disorder. To target levels of clutter, the investigators are testing an intervention to add in-home decluttering practice to the BIT workshop.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at consent
* Primary hoarding disorder, Saving Inventory Revised greater than or equal to 40.
* Clutter Image Rating Scale greater than or equal to 3 and less than or equal to 7.
* Low risk for eviction
* English speaking
* Will and able to understand and complete consent procedures

Exclusion Criteria:

* Hoarding disorder not primary
* Severely depressed individuals; Hamilton Depressions Rating Scale greater than 30 or judged clinically to be at risk of suicide with Columbia Suicide Severity Scale
* Unable or unwilling to allow study staff into home for home assessment OR a Clutter Image Rating Score of less than 2 or greater than 7.
* At risk for eviction
* Animal Hoarding or squalor of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Blair Simpson, MD, PhD, Principal Investigator — Columbia-NYSPI-RFMH

REFERENCES:
- [Result] Linkovski O, Zwerling J, Cordell E, Sonnenfeld D, Willis H, La Lima CN, Baker C, Ghazzaoui R, Girson R, Sanchez C, Wright B, Alford M, Varias A, Filippou-Frye M, Shen H, Jo B, Shuer L, Frost RO, Rodriguez CI. Augmenting Buried in Treasures with in-home uncluttering practice: Pilot study in hoarding disorder. J Psychiatr Res. 2018 Dec;107:145-150. doi: 10.1016/j.jpsychires.2018.10.001. Epub 2018 Oct 5. PMID 30419524

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not applicable. Participants did not have a wash out or run-in.
Period: Overall Study
Arm/Group | Experimental: BIT+In-home Decluttering
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: BIT+In-home Decluttering
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Savings Inventory Revised
Description: The Saving Inventory-Revised scale (SI-R) is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.
  The total score (sum of 23 items) ranges from 0 to 92. Total score higher than 41 shows significant difficulty with clutter.
  For the acquisition subscale we sum items 2 (reverse score), 9, 11, 14, 16, 18 and 21. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with excessive acquisition.
  For the difficulty discarding subscale we sum items 4(reverse score), 6, 7, 13, 17, 19, 23. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with discarding.
  For the clutter subscale we sum items 1, 3, 5, 8, 10, 12, 15, 20, 22. The subscale ranges from 0 to 36 and score greater than 15 indicates difficulty with accumulated clutter.
Time Frame: Change from baseline at 0, 12 weeks and 18 weeks after treatment start
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Experimental: BIT+In-home Decluttering
Number analyzed (Participants) | 5
units on a scale
  Baseline | 71 [62 to 75]
  12 weeks | 55 [45 to 70]
  18 weeks | 53 [23 to 66]

2. Primary Outcome: Clutter Image Rating Scale
Description: Three sets of photographs, each containing nine photos of a single room with varying levels of clutter. A selection is made as to which photograph best resembles their own home.
  This scale assesses the clutter levels in the bedroom, living room and kitchen. The scale for each room ranges from 1 to 9. Clutter that reaches the level 4 indicates significant difficulty with clutter that affects the person's life.
Time Frame: Change from baseline at 0, 12 weeks and 18 weeks after treatment start
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Experimental: BIT+In-home Decluttering
Number analyzed (Participants) | 5
units on a scale
  Baseline | 4.7 [4.0 to 7.0]
  12 weeks | 4.7 [2.7 to 4.7]
  18 weeks | 2.7 [1.0 to 6.3]

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: No adverse events reported by participants
Arm/Group | Experimental: BIT+In-home Decluttering
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes